CLINICAL TRIAL: NCT03150758
Title: Intra-operative Assessment of Cavernosal Nerve Stimulus Threshold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE1816
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Results first posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Prostatectomy
Keywords: Erectile Disfunction; Urinary Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Electrical Stimulation (Experimental): Each participant will be given 4 electrical stimulants with an amplitude ranging from 1mA to 30mA. The maximum stimulus without causing an erection will be recorded
  Interventions: Device: 10Hz + 100 micro-seconds; Device: 10Hz + 200 micro-seconds; Device: 7Hz + 100 micro-seconds; Device: 7Hz + 200 micro-seconds

INTERVENTIONS:
Device: 10Hz + 100 micro-seconds — 10Hz Electrical Stimulation with a pulse width of 100 micro-seconds
Device: 10Hz + 200 micro-seconds — 10Hz Electrical Stimulation with a pulse width of 200 micro-seconds
Device: 7Hz + 100 micro-seconds — 7Hz Electrical Stimulation with a pulse width of 100 micro-seconds
Device: 7Hz + 200 micro-seconds — 7Hz Electrical Stimulation with a pulse width of 200 micro-seconds

SUMMARY:
Erectile dysfunction persists in approximately 80% of men 1 year after prostatectomy. Various erectile rehabilitation strategies have not provided benefit. Electrical stimulation has been demonstrated to benefit neuroregeneration and the functional recovery of neuromuscular systems. Therefore, electrical stimulation of the cavernosal nerves during radical prostatectomy is being investigated for its potential development into a treatment aimed at improving recovery of erectile function after prostatectomy. This pilot study is intended to determine the threshold of electrical stimulation that results in penile erection, as defined by persistent intracavernosal pressure increase, such that future studies of sub-threshold stimulation may be pursued.

DETAILED DESCRIPTION:
Objective:

To determine the cavernosal nerve electrical stimulation amplitude thresholds at which an erection, as indicated by persistent increases in intracavernosal pressure, occurs for various stimuli of fixed frequency and fixed pulse-width.

Study Design:

This is a prospective pilot study used to determine a threshold range of cavernosal nerve electrical stimulation parameters that result in penile erection. Assignment to the order of stimulation paradigms will be randomized. No placebos are used. No blinding is used.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have prostate cancer being treated via radical prostatectomy by a single surgeon (primary investigator) with planned intraoperative nerve sparing.
* Subjects must have intact preoperative erectile function, sufficient for penetrative intercourse without medication nor assistive device, as defined by a Sexual Health Inventory for Men (SHIM) / International Index of Erectile Function (IIEF-2) score 22 or higher, which is collected as part of routine care.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Baseline erectile dysfunction, as defined by the use of medications or devices to assist erection, lack of baseline erections, or a SHIM / IIEF-2 21 or lower, which is collected as part of routine care.
* Lack of successful intraoperative nerve sparing.
* Neurologic, metabolic, or vascular diseases that may negatively impact erectile function, such as: diabetes mellitus, peripheral vascular disease, coronary artery disease, stroke, multiple sclerosis, parkinson's disease, multiple systems atrophy, epilepsy, or spinal cord injury.
* Inability to provide a fully informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Klein, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Electrical Stimulation
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who were put on study
Arm/Group | Electrical Stimulation
Number analyzed (Participants) | 6
Age, Customized [Number; unit: participants]
  20-29 years | 0
  30-39 years | 0
  40-49 years | 0
  50-59 years | 6
  60-69 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Cavernosal Nerve Stimulation Threshold
Description: Median value of "maximum stimulation pattern men received prior to erection" in responders
Time Frame: Up to 21 days after prostatectomy
Population: Participants who responded to therapy
Measure: Median (Inter-Quartile Range); unit: mA
Arm/Group | Electrical Stimulation
Number analyzed (Participants) | 6
mA | 7.5 [5 to 11.25]

ADVERSE EVENTS:
Time Frame: up to 30 days from end of treatment
Arm/Group | Electrical Stimulation
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-03-29): https://cdn.clinicaltrials.gov/large-docs/58/NCT03150758/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT03150758/ICF_001.pdf